CLINICAL TRIAL: NCT01888042
Title: Phase II Study Assessing Everolimus as Fist Line Treatment in Patients With Metastatic Kidney Cancer of Bad Prognosis
Brief Title: Assessing Everolimus in Fist Line Treatment on Patients With Metastatic Kidney Cancer
Acronym: POORTOR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-00979-14; 2011/1733 (Other: CSET number)
Record Dates: First submitted 2013-06-25; First posted 2013-06-27 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Kidney Cancer
MeSH Terms: conditions — Kidney Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Everolimus (Experimental): Everolimus will be administered per os every day at the same hour immediately after a meal with a glass of water 10 mg (1 tablet of 10 mg)
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — 10 mg (1 tablet of 10 mg)

SUMMARY:
It is a an open label, multicentric, phase II study assessing the efficacy of everolimus (given per os) as a first line treatment in kidney cancer of bad prognosis.

92 patients will be included (anticipated). The treatment by everolimus will continue until progression, significant toxicity or withdraw of consent

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic kidney cancer, regardless of histology (except Bellini carcinomas), with measurable or evaluable disease
2. Age >= 18 years
3. With Karnofsky ≥ 60
4. Without prior treatment for metastatic cancer (chemotherapy, targeted therapy, or mTOR inhibitor)
5. Bad prognosis, defined as follows: at least three of the following six criteria of poor prognosis:

   * Karnofsky <80
   * LDH> 1.5 ULN
   * hemoglobin <LLN
   * corrected calcium> 2.5 mmol / l (10 mg / dl)
   * Time frame between initial diagnostic and treatment <1 year
   * More than one metastatic site
6. medullary function: neutrophils ≥ 1.5 x 109 / L, Platelets ≥ 100 x 109 / L, Hb> 8g/dL
7. Hepatic function: bilirubin: ≤ 1.5 x ULN, ALT and AST ≤ 2.5x ULN in the absence of hepatic metastasis ≤ 5x ULN if hepatic metastasis documented
8. Renal function: creatinine <1.5 x ULN
9. Life expectancy> 3 months,
10. Patient signed informed consent and agreeing to comply with the requirements of the trial

Exclusion Criteria:

1. Previous treatment with chemotherapy, targeted therapy, or mTOR inhibitor
2. Previous radiotherapy in the last 2 weeks
3. Chronic treatment with corticoids or immunosuppressive agents except substitutive opotherapy.. A washout period of at least 8 days must be respected before the patient inclusion.
4. Patients with brain metastases untreated or uncontrolled by prior treatment. The non-progression of the metastases must be proved by comparing two brain scans separated by a minimum interval of 6 weeks.
5. Active bleeding
6. Patient with positive serology HBs (Ag HBs (+) and AC anti-HBc (+)
7. Hypersensitivity to everolimus, sirolimus, to other rapamycin derivatives or to any of the excipients
8. Severe or uncontrolled medical pathology:

   * unstable angina, symptomatic heart failure, myocardial infarction ≤ 6 months before randomization, severe rhythm disorder,
   * Uncontrolled diabetes with glycaemia> 1.5X ULN.
   * Active or uncontrolled infection.
   * cirrhosis or chronic active hepatitis,
   * severe alteration in lung function (> 50% decrease in FEV or vital capacity)
9. Other cancer within the past 3 years, with the exception of basal cell carcinoma and carcinoma in situ of the cervix
10. Pregnant or lactating woman, and adults refusing an effective contraceptive method
11. Participation in another clinical trial with an investigational drug
12. Refusal of the patient to comply with the rules of the clinical trial
13. Person deprived of liberty or person under guardianship, inability to submit to medical treatment test for geographical, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | From inclusion to progression, significant toxicity or death wichever come first up to 56 months

SECONDARY OUTCOMES:
Response rate | From inclusion to progression, significant toxicity or death whichever come first up to 56 months
  Response rate based on RECIST 1.1 criteria
Toxicity of Everolimus | From inclusion to progression, significant toxicity or death whichever come first up to 56 months
Progression Free Survival (PFS) | From inclusion to progression, significant toxicity or death whichever come first up to 56 months

CONTACTS AND LOCATIONS:
Overall Officials: Bernard ESCUDIER, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Gustave Roussy, Villejuif, Val de Marne, France